CLINICAL TRIAL: NCT07326475
Title: Comparison of Selected Physiotherapeutic Interventions on Kinetic and Kinematic Parameters in Young Soccer Players
Brief Title: Comparison Interventions on Kinetic and Kinematic Parameters
Acronym: Balance
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: KB/523/2025
Record Dates: First submitted 2025-11-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Young Football Players; Ankle Sprain Prevention
Keywords: soccer; proprioception; manualn therapy; postural balance; biomechanics
MeSH Terms: interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A "Diagonal Mobilization' (Experimental): Will be used: manipulation, placebo and exercise
  Interventions: Other: Manual therapy; Other: Placebo; Other: Exercise
- Group B "Placebo" (Placebo Comparator): Will be used: manipulation, placebo and exercise
  Interventions: Other: Manual therapy; Other: Placebo; Other: Exercise
- Group C "Proprioception Training" (Active Comparator): Will be used: manipulation, placebo and exercise
  Interventions: Other: Manual therapy; Other: Placebo; Other: Exercise

INTERVENTIONS:
Other: Manual therapy — This technique involves mobilizing the upper ankle joints by mobilizing the talus and calcaneus, improving pronation.
Other: Placebo — The players will perform their own type of pro-receptive training.
Other: Exercise — Pro-receptive training will be performed.

SUMMARY:
Currently, it is difficult to find studies in the literature comparing proprioception exercises with the effect of manual therapy on improving balance, and in the long run it may translate into improved activity, functionality and injury prevention in athletes, when planning training or therapy, e.g. in patients after ankle sprains.

ELIGIBILITY:
Inclusion Criteria:

* Age 11-13 years
* Male
* Minimum 2 years of experience in soccer coaching
* Participation in regular club training (at least 3 times a week)
* Parental/legal guardian consent and participant consent to participate in the study
* No medical contraindications to physical activity

Exclusion Criteria:

* Current injury or contusion of the musculoskeletal system that prevents full participation in training
* Chronic diseases that may affect the musculoskeletal system or balance
* Participation in other training programs focused on proprioception or undergoing other physiotherapy interventions during the study period

Ages: 11 Years to 13 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 45 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Y balance test | The test will be administered twice during a single training session. Baseline (0 minutes before the intervention) and immediately post-intervention (within 5 minutes after completion of the training session). Each test will be repeated three times.
  Consists of the volunteer standing on one leg while simultaneously stretching the other lower limb in 3 different directions. These are: anterior, posteromedial and posterolateral.
1. Balance | The test will be administered twice during a single training session. Baseline (0 minutes before the intervention) and immediately post-intervention (within 5 minutes after completion of the training session). Each test will be repeated three times.
  K-FORCE plates assess balance characteristics during testing.

SECONDARY OUTCOMES:
Assessment of proprioception. | The test will be administered twice during a single training session. Baseline (0 minutes before the intervention) and immediately post-intervention (within 5 minutes after completion of the training session). Each test will be repeated three times.
  The proprioception assessment involves assessing the angular position of the joint and then attempting to reproduce it, measured in degrees. The assessment will be conducted at 30 degrees, 60 degrees, and 90 degrees.
Muscle strength assessment | The test will be administered twice during a single training session. Baseline (0 minutes before the intervention) and immediately post-intervention (within 5 minutes after completion of the training session). Each test will be repeated three times.
  The K-FORCE Push Test allows you to assess your strength characteristics during the hip abduction test.

CONTACTS AND LOCATIONS:
Locations (1):
- Escola Futbolu Pruszcz Gdański, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No